CLINICAL TRIAL: NCT01527227
Title: Parentification Among Children Whose Parents Cope With a Serious Mental Illness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 84-11
Record Dates: First submitted 2011-11-21; First posted 2012-02-06 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-01

CONDITIONS: Mental Illness
Keywords: Children of mentally ill
MeSH Terms: conditions — Mental Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children of mentally ill: This research will include 130 children between the ages of 10-18 who live with at least one parent who struggles with serious mental illness in a comparison to 130 children of the same socio-demographic characteristics raised by parents from a non-clinical population
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — The research will examine effects of personal, familial, societal and intergenerational characteristics on parentification, the effects of parentification on the quality of life of the child and what encourages a better quality of life.

SUMMARY:
The research will examine effects of personal, familial, societal and intergenerational characteristics on parentification, the effects of parentification on the quality of life of the child and what encourages a better quality of life. This research will include 130 children between the ages of 10-18 who live with at least one parent who struggles with serious mental illness in a comparison to 130 children of the same socio-demographic characteristics raised by parents from a non-clinical population. The differences between these two populations with regard to parentification, quality of life, social support and fairness will also be examined. The parents and the children will fill out questionnaires. The research group will be recruited from rehabilitation services, mental health clinics, psychiatric hospitals and social welfare departments with sampling method. The comparison group will be recruited from schools. This research broadens the knowledge of the causes and the repercussions of parentification among children of parents who struggles with serious mental illness in comparison with children raised by parents from a non-clinical population. Few studies have examined children of the mentally ill in Israel, and there are none which examined parentification.

ELIGIBILITY:
Inclusion Criteria:

* children who live with at least one parent who struggles with serious mental illness

Exclusion Criteria:

* Arabic children

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The research group will be recruited by the WHO and ICMJE with sampling method. The comparison group will be recruited from schools.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Filial Responsibility Scale-Youth (child fill out) | 1 year
  Responses to the 34-items are given on a 4-point Likert scale ("not at all true" to "very true") and assess instrumental caregiving (e.g., "I work to make money for my family"),emotional caregiving (e.g., "I often try to keep the peace in my family")and perceived fairness (e.g., "In my family, I am often asked to do more than my share."). Higher scores indicate higher levels of caregiving and perceived fairness.

SECONDARY OUTCOMES:
The Social Support Appraisals Scale (Dubow & Ullman,1989)(child fill out) | 1 year
  31-item scale assesses the child's appraisals of peer, family, and teacher support.The child responds to each item on a 5-point continuum (1 = always, 5 =never).
"The Alabama Parenting Questionnaire"; Shelton, Frick & Wootton, 1996 (parent fill out) | 1 year
  The APQ measures five dimensions of parenting that are relevant to the etiology and treatment of child externalizing problems: (1) positive involvement with children, (2) supervision and monitoring, (3) use of positive discipline techniques, (4) consistency in the use of such discipline and (5) use of corporal punishment.
  This study use only positive involvement dimension
Parental Bonding Instrument (PBI) (parent fill out) | 1 year
  Two scales termed 'care' and 'overprotection' or 'control', measure fundamental parental styles as perceived by the child. The measure is 'retrospective', meaning that adults (over 16 years) complete the measure for how they remember their parents during their first 16 years. The measure is to be completed for both mothers and fathers separately. There are 25 item questions, including 12 'care' items and 13 'overprotection' items.
Social support and social conflict (parent fill out) | 1 year
  Questions were developed to measure the affect, affirmation, and aid components of social support from Extended family and spouse. social support and social conflict items were rated on 5-point Likert-type scales with options that ranged from not at all to a great deal

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Services, All the Country, Israel, Israel